CLINICAL TRIAL: NCT03554733
Title: A Bridge From Rehabilitation to Real-World: Re-Inventing Yourself After SCI
Brief Title: Bridge Reinvention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Coker, Research Associate, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2959
Record Dates: First submitted 2018-05-30; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Spinal Cord Injuries
Keywords: self efficacy; participation; satisfaction with life
MeSH Terms: conditions — Spinal Cord Injuries; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Single-blind, waitlist-control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Re-Inventing Yourself after SCI protocol - 6-week educational sessions
  Interventions: Behavioral: ReInventing Yourself after SCI
- Control (No Intervention): No intervention during course of study; participants offered the option of receiving the study intervention after completion of study.

INTERVENTIONS:
Behavioral: ReInventing Yourself after SCI — 6-week, manualized, cognitive-behaviorally based group educational intervention
  Arms: Treatment

SUMMARY:
The goal of this randomized controlled trial is to determine the efficacy of a treatment to improve resilience to stress for individuals with SCI who are transitioning from inpatient rehabilitation to home. The overarching hypothesis is that individuals who participate in an intervention that presents positive psychotherapy topics in an interactive, structured, cognitive-behaviorally-based group intervention that stresses restructuring maladaptive thought processes and provides experiential opportunities to reinforce behavioral change will demonstrate increased self-efficacy.

DETAILED DESCRIPTION:
The goal of this randomized controlled trial is to determine the efficacy of a treatment to improve resilience to stress for individuals with SCI who are transitioning from inpatient rehabilitation to home. The overarching hypothesis is that individuals who participate in an intervention that presents positive psychotherapy topics in an interactive, structured, cognitive-behaviorally-based group intervention that stresses restructuring maladaptive thought processes and provides experiential opportunities to reinforce behavioral change will demonstrate increased self-efficacy. There were three aims of this study: AIM 1: Self-Efficacy - To examine the ability of a six-week, manualized, cognitive-behaviorally based group educational intervention (Re-Inventing Yourself after SCI-Bridge) to improve both SCI-specific and general self-efficacy for people who are early in the process of community reintegration; AIM 2: Psychosocial Adjustment - To assess the ability of the Re-Inventing Yourself after SCI-Bridge intervention to improve psychosocial adjustment of people with SCI who are early in the community reintegration process; and, Aim 3: Participation - To determine the ability of the Re-Inventing Yourself after SCI-Bridge intervention to improve societal participation for people with SCI who are early in the community reintegration process.

ELIGIBILITY:
Inclusion Criteria:

1. History of SCI at any level;
2. completed initial inpatient rehabilitation but are no more than 6 months post-discharge;
3. 18 years of age or older at the time of study enrollment;
4. English speaking in order to complete study measures and participate in group interactions; and
5. able to provide informed consent to participate.

Exclusion Criteria:

1. History of moderate or severe traumatic brain injury;
2. current participation in another RCT;
3. live beyond a reasonable commuting distance from Craig Hospital;
4. unable to verbally communicate;
5. unable to attend group sessions;
6. active participation in another formal clinical group or psychological therapy;
7. are currently experiencing severe depression which would require more intense treatment than is provided in this intervention, as evidenced by a score of 20 or higher on the Personal Health Questionnaire-9;
8. report any current suicidal ideation on the Personal Health Questionnaire-9; or
9. have any condition that, in the judgment of the investigators, precludes successful participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Moorong Self-Efficacy Scale (MSES) | Baseline, 6 weeks, 12 weeks, 18 weeks
  The MSES is a 16 item self-report measure of self-efficacy related to everyday life activities, designed specifically for persons with SCI. Individuals use a 7-point Likert scale ranging from 1 (very uncertain) to 7 (very certain) to rate their ability to perform 16 everyday tasks, with higher scores representing greater perceived self-efficacy. A Total Score, ranging from 16 to 112 is calculated by summing all item responses. The MSES has been used in previous studies of SCI, and demonstrates excellent internal consistency (alpha = 0.91 - 0.93), high reliability, and good convergent, concurrent and divergent validity. Time to administer: 5 to 10 minutes.

SECONDARY OUTCOMES:
Change in Generalized Self-Efficacy Scale (GSES) | Baseline, 6 weeks, 12 weeks, 18 weeks
  The GSES is a questionnaire designed to assess a person's ability to cope with a variety of difficult demands in life, with ten items scored using a Likert rating scale, ranging from 1 (not at all true) to 4 (exactly true). This scale has acceptable internal reliability (ranging from.73 to .90) and criterion validity, as demonstrated by positive correlations with positive emotions, optimism, and work satisfaction, and negative correlations with anxiety, stress, depression, and health complaints. The GSES has been used and validated in numerous populations and cultures, including people with SCI. This self-administered scale produces a Total Score ranging from 10-40, with higher scores indicating greater general self-efficacy. Time to administer: 3 to 5 minutes.
Change in Satisfaction with Life Scale (SWLS) | Baseline, 6 weeks, 12 weeks, 18 weeks
  The SWLS is a five item measure on which respondents rate their life satisfaction using a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree). A Total Score is calculated by summing each of the items, having a range of 5 to 35, with higher scores representing greater perceived quality of life. This measure has well established psychometric properties, with high reliability (.79 to .89), good content validity, criterion validity, and has been extensively used in research regarding people with SCI. Time to administer: 1 to 3 minutes.
Change in Participation Assessment with Recombined Tools - Objective (PART-O) | Baseline, 6 weeks, 12 weeks, 18 weeks
  The PART-O is a 17-item assessment of participation and has demonstrated good psychometric properties in measuring participation for people living with disabilities. The PART-O has acceptable reliability and validity for persons with SCI. An Averaged Total Score is computed by taking the mean of 17 items, with scores ranging from 0 (never participate in these types of activities) to 5 (almost always participate in these types of activities), with higher scores representing greater participation. This assessment will be utilized to measure overall participation. Time to administer: 8 to 10 minutes.
Patient Health Questionnaire - 9 (PHQ-9) | Baseline, 6 weeks, 12 weeks, 18 weeks
  The PHQ-9 is a 9 item scale that will be used to assess depression. Respondents rate the frequency at which specific problems have been bothersome during the past two weeks, using a four point scale ranging from 0 (not at all) to 3 (nearly every day). A total score is calculated by summing all items, with higher scores indicating an increasing severity of depression. This scale demonstrates excellent psychometrics, with excellent internal consistency (α = 0.86 - 0.89), high test-retest reliability (0.84) and good criterion and construct validity and has been used extensively in populations with SCI. Time to administer: 1 to 3 minutes.
Change in General Anxiety Disorder 7-item (GAD-7) | Baseline, 6 weeks, 12 weeks, 18 weeks
  The GAD-7 is a brief 7 item measure that will be used to assess the severity of general anxiety. Using a four point Likert scale ranging from 0 (not at all sure) to 3 (nearly every day), respondents rate how often they have been bothered by specific symptoms during the past two weeks. A total severity score, ranging from 0 to 21, is calculated by summing all items. This measure has demonstrated high internal consistency (α = .89 - .92), good test-retest reliability (icc = .83) and adequate convergent and discriminant validity. This scale has been used in previous studies involving persons with SCI. Time to administer: 1 to 3 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Coker, MPH, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No